CLINICAL TRIAL: NCT05627648
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Parallel-Group Confirmatory Study For Intracordal Administration Of KP-100LI In Patients With Vocal Fold Scar
Brief Title: Phase 3 Study of KP-100LI in Subjects With Vocal Fold Scar
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kringle Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KP-100-FD001
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Vocal Fold Scar
Keywords: Hepatocyte Growth Factor; HGF; KP-100LI; KP-100; intracordal injection
MeSH Terms: conditions — Deafness, Autosomal Recessive 39 | interventions — Hepatocyte Growth Factor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KP-100LI (Active Comparator): Intracordal injection, 20 mcg once per week, 3 weeks
  Interventions: Drug: KP-100LI
- Placebo (Placebo Comparator): Intracordal injection, once per week, 3 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KP-100LI — Intracordal injection, 20 mcg once per week, 3 weeks
  Other Names: Hepatocyte Growth Factor; HGF
  Arms: KP-100LI
Drug: Placebo — Intracordal injection, once per week, 3 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm the efficacy and safety of KP-100LI, a intracordal formulation containing recombinant human dHGF as the active pharmaceutical ingredient, for voice function improvement therapy in patients with vocal fold scar (including vocal fold sulcus).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years to 75 years
2. Presence of bilateral vocal fold scar or sulcus diagnosed
3. No other vocal lesion or vocal movement disorder
4. Voice Handicap Index-10 (VHI-10) score of 11 or higher
5. No laryngoplasty, collagen or lipid infusion to vocal cord, removal scar, fascial graft, or administration of steroid or hyaluronic acid to vocal cord

Exclusion Criteria:

1. No movement disorders of the vocal fold including paralysis
2. Airway disease caused by burn
3. History of malignant tumor
4. History of allergy to local anesthesia agent
5. With impaired coagulation-fibrinolysis, or taking anticoagulant or antiplatelet drugs
6. Serious concomitant disease
7. Pregnant (including suspected), nursing, wishing to become pregnant, or unable to prevent conception during the trial period using contraceptive methods

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Improvement rate in Voice Handicap Index-10 (VHI-10) score at 24 weeks of the observational period | 24 weeks

SECONDARY OUTCOMES:
Improvement rate in VHI-10 score from just before the first administration ("baseline" at 0 week) to 4, 8, and 12 weeks of the observational period | up to 12 weeks
Changes in VHI-10 score from baseline to 4, 8, 12, and 24 weeks of the observational period | up to 24 weeks
Changes in Normalized Mucosal Wave Amplitude (NMWA) from baseline to on 4, 8, 12, and 24 weeks of the observational period | up to 24 weeks
Changes in GRBAS (Grade, Roughness, Breathiness, Asthenia, Strain) scale from baseline to on 4, 8, 12, and 24 weeks of the observational period | up to 24 weeks
Evaluation of adverse events | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daichika Hayata, Study Director — Kringle Pharma, Inc.
Locations (8):
- Japan (8):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Fukuoka Sanno Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - University Hospital Kyoto Prefectural University of Medicine, Kamigyō-ku, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Kawasaki Medical School Hospital, Kurashiki, Okayama-ken
  - Nihon University Hospital, Chiyoda-ku, Tokyo
  - Sanno Medical Center, Minato-Ku, Tokyo